CLINICAL TRIAL: NCT02996721
Title: A Trial Evaluating Vitamin D Normalization on Major Adverse Cardiovascular-Related Events Among Myocardial Infarction Patients (The TARGET-D Study)
Brief Title: A Trial Evaluating Vitamin D Normalization on Major Adverse Cardiovascular-Related Events Among Myocardial Infarction Patients
Acronym: TARGET-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1050296
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Death; Myocardial Infarction; Cerebral Vascular Accident; Heart Failure Hospitalization
MeSH Terms: conditions — Death; Myocardial Infarction; Stroke | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients randomized to the standard of care arm will have a 25[OH] Vit D test performed, a sample taken and stored for future tests, and completion of a PHQ-9 depression survey at baseline and at study conclusion. No other contact is planned with the standard of care patients. Follow-up will be done by the querying of electronic records, which includes any 25[OH] Vit D testing, use of vitamin D supplementation, and outcomes.
- Treatment (Experimental): Patients randomized to the treatment arm will have a 25[OH] Vit D test performed, a sample taken and stored for future tests, and completion of a PHQ-9 depression survey. If at baseline a patient has a 25[OH] Vit D >40 ng/mL then follow-up testing will occur 1 year from baseline and the patient will continue current treatment strategy (no supplementation or current supplementation dosage). If baseline 25[OH] Vit D levels are <40 ng/mL then the patient will initiate or increase dose and return in 3 months (±15 days) to determine 25[OH] Vit D level. At 3 months, if 25[OH] Vit D >40 ng/mL then current dose should be kept and the patient will return in 1 year for follow-up testing. However, if 25[OH] Vit D <40 ng/mL then patients should double current dose and test again in 3 months. This should occur until 25[OH] Vit D reaches a level >40 ng/mL and once achieved, the patient will return in 1 year for follow-up 25[OH] Vit D testing.
  Interventions: Biological: Vitamin D3

INTERVENTIONS:
Biological: Vitamin D3 — Vitamin D3 (cholecalciferol) will be provided to participants of the study.
  Arms: Treatment

SUMMARY:
This study evaluates whether achieving 25-hydroxyvitamin D (25[OH] Vit D) levels (>40 ng/mL) among myocardial infarction patients will result in a reduction of cardiovascular-related adverse events. Half of the patients will be randomized to receive standard of care and half will receive clinical management of 25[OH] Vit D levels.

DETAILED DESCRIPTION:
Low 25[OH] Vit D levels have become a public epidemic with increasing recognition of its widespread insufficiency both in the United States and worldwide. Epidemiologic studies have associated low 25[OH] Vit D levels with coronary risk factors and adverse cardiovascular outcomes. However, randomized trials are needed to establish the relevance of 25[OH] Vit D status to cardiovascular health. While a few randomized trials have evaluated vitamin D supplementation, none have "treated to target" (i.e., individual dosing so that adequate 25[OH] Vit D levels are obtained), but have rather given "blanket" doses regardless of 25[OH] Vit D level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, both male and female, >18 years old
2. Undergone angiography for a MI (troponin positive [>0.04 ng/mL] and ACS diagnosis) within the past month
3. Receive follow-up care at an Intermountain Healthcare facility
4. Not taking or taking <1000 IU of vitamin D daily within the last 3 months
5. Willing to provide informed consent and participate in follow-up visits

Exclusion Criteria:

1. Hypersensitivity to vitamin D products
2. History of previous vitamin D supplementation of >1000 IU daily within the past 3 months (i.e., >40% of the days during the past 3 months).
3. Systemic disease (including terminal cancer, cirrhosis, end stage COPD, etc) with a reduced (<12 months) life expectancy
4. Hypercalcemia (calcium levels >10.6 mg/dL)
5. Subject participation in previous investigational interventional studies within 30 days of the current study.
6. History of psychiatric illness/condition that would interfere with their ability to understand or complete the requirements of the study, a condition that in the opinion of the investigator or their designee places the subject at an unacceptable risk as a participant.
7. Pregnant and/or lactating women and women of child bearing potential who are not using acceptable means of contraception as determined by the clinical investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Composite Outcome of Death, Myocardial Infarction, Heart Failure Hospitalization, and Cerebral Vascular Accident | from date of randomization until the date of first documented event, up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi T May, PhD, MSPH, Principal Investigator — Intermountain Heart Institute; Joseph B Muhlestein, MD, Principal Investigator — Intermountain Heart Institute
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No